CLINICAL TRIAL: NCT03757468
Title: Pain and Discomfort During Maxillary Expansion: A Randomized Multicentric Study
Brief Title: Pain and Discomfort During Maxillary Expansion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Genova (Other)
Collaborators: University of Milan (Other)
Responsible Party: Principal Investigator, ALESSANDRO UGOLINI, Assistant Professor, University of Genova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCT_Milano-Genova
Record Dates: First submitted 2018-11-12; First posted 2018-11-29 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Crossbite; Maxillary Hypoplasia
MeSH Terms: conditions — Malocclusion; Retrognathia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RME (rapid maxillary expander) (Active Comparator): Intervention orthodontic - maxillary expansion : crossbite or transversal maxillary deficiency correction with the standard hyrax expansion screw anchored on second deciduous molars
  Interventions: Device: orthodontic - maxillary expansion
- Leaf (leaf maxillary expander) (Experimental): Intervention orthodontic - maxillary expansion : crossbite or transversal maxillary deficiency correction with Leaf Expander appliance anchored on second deciduous molars.
  Interventions: Device: orthodontic - maxillary expansion

INTERVENTIONS:
Device: orthodontic - maxillary expansion — After appliance placement, the screw (hyrax or leaf type) will be activated until overcorrection. Expansion will be considered adequate when the occlusal surface of the first maxillary palatal cusp contact the occlusal surface of the mandibular first molar facial cusp. When will be achieved, the expander will stay in place for 10 months.
  Other Names: orthodontic - palatal expansion

SUMMARY:
The aim of the present study is to investigate and analyze the perception of pain and function impairment during the first week of activation with two different palatal expansion screw to identify an effective pain prevention protocol.

DETAILED DESCRIPTION:
Maxillary expansion with fixed appliance is a well-known and consolidated practice in clinical orthodontics but current findings of "evidence based dentistry" have not yet identified a better clinical expansion protocol. This issue is due both to the several expansion screws available on the market and to the different screw activation protocols, which could be grouped into rapid and slow, with several customizations. A recent systematic review has shown that both rapid and slow expansion protocols are clinically effective on the primary outcome, i.e. the resolution of the crossbite with a significant increase of skeletal transversal dimension in the maxillary transverse deficiency subjects. If the type of appliance based on its ability to solve the maxillary constriction is not any more the main selection criteria, the choice of the orthodontist should, therefore, be based on the timing and on a "patient-oriented" device, that minimizes the side effects, such as e.g. appliance breakages, functional impairments and pain.

In the orthodontic daily practice, the pain of the little patient is the most frequent symptom during treatment and is the one that most frightens/worries the child and the family. Literature shows that rapid maxillary expansion is, among the early orthodontic therapies, the one with the highest frequency of pain (up to 98%) as an adverse symptom reported by patients. The pain is statistically linked to the rapid expansion protocol (2/turn/day), during which, for each activation of the screw (0.2 or 0.25 mm) the force expressed can reach up to 10 pounds which acts in an orthopaedic manner on the palatine suture and the circummascellar sutures. Following this orthopedic action, a disorganized and highly vascularized connective tissue (inflammatory) is formed in palatine suture area, which becomes the main receptor of the pain perceived by the patient during the active maxillary expansion. In the literature the prevention and management of pain during palate expansion is a poorly analyzed topic, despite being a daily problem in orthodontic clinical practice and so the aim of the present study is to investigate and analyze the perception of pain and function impairment during the first week of activation with two different palatal expansion screw to identify an effective pain prevention protocol.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with transversal maxillary deficiency (with or without crossbite).
* Class I or Class II dental malocclusion with uni- or bilateral crossbite and/or constricted maxilla
* Before the pubertal peak (CVM 1-3).

Exclusion Criteria:

* Patients with previous orthodontic treatment
* Hypodontia in any quadrant excluding third molars
* Inadequate oral hygiene
* Craniofacial syndromes, or cleft lip or palate

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-07-30 (Estimated); Study Completion 2019-07-30 (Estimated)

PRIMARY OUTCOMES:
Crossbite correction | 10 months
  Clinical evaluation in vivo (binary outcome yes/no)
Traversal maxillary deficiency correction | 10 months
  Measured on digital dental casts (increase in mm of the intermolar and intercanine width)
Pain during active expansion phase | 1 week
  Pain reported on Wong-Baker Faces Pain Scale analysis. Pain intensity was assessed using the Wong-Baker scale (Wong and Baker, 1988) from the first to the seventh day of the screw activation, reporting a daily registration in the evening. The Wong-Baker scale is a tool for self-assessment of pain intensity and is used in children from three years of age. The smiles range from the most smiling, corresponding to "no pain", to the one that cries, corresponding to "worst pain imaginable". Each face is also paired with a number, from 0 to 10, which coincides with the intensity of the pain. Higher values represent a worse outcome.
Discomfort during active expansion phase | 1 week
  Discomfort reported on a questionnaire

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Università di Genova, Genova, GE
  - Università di Milano, Milan

IPD SHARING:
Plan to Share IPD: No